CLINICAL TRIAL: NCT06194058
Title: Rapid Sequence Intubation and Hemodynamic Disorders in the Operating Room: a Prospective Multicenter Observational Study. The Crush or Crash Study.
Brief Title: Rapid Sequence Intubation and Hemodynamic Disorders in the Operating Room: a Prospective Multicenter Observational Study
Acronym: CoC
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: AR_2023_001
Record Dates: First submitted 2023-11-14; First posted 2024-01-08 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Rapid Sequence Intubation
Keywords: anesthetic induction; adult patients; hemodynamic disorders; arrythmia; cardiac arrest; pre-oxygenation; mean blood pressure
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: rapid sequence anesthetic induction — Rapid sequence induction and intubation (or crash induction) is a process for inducing general anesthesia when the patient is at a high risk of pulmonary aspiration. It aims at minimizing the time between giving the induction drugs and securing the tube, during which period the patient's airway is essentially unprotected.

SUMMARY:
There is a great heterogeneity in the practice of rapid sequence induction in the operating room in the world. There are no recent data assessing the rate of implementation of the latest French formalized expert recommendations in clinical practice. In addition, the modalities for the management of haemodynamic disorders, particularly hypotensive disorders, during rapid sequence induction are not described in these recommendations, although these are frequent events with a non-zero morbidity mortality potential.

The goal of this prospective, observational, multicenter, anesthetic study is to describe the clinical practice of French anesthesiologists regarding the prevention of severe hemodynamic disorders during rapid sequence anesthetic induction in adult patients.

The primary outcome measure is the occurrence of a major haemodynamic disorder defined by a MBP ≤ 50 mmHg (or ≤ 40% of the reference value) and/or ≥ 110 mmHg and/or the occurrence of sustained arrhythmia not present at induction and/or cardiac arrest within the first 10 minutes after induction of anesthesia.

The clinical practices of pre-oxygenation, induction and intubation of French anesthesiologists and compliance with the formalized expert recommendations of 2017 and 2018 will also be studied secondarily. The elements for the prevention of gastric fluid inhalation, the organization and equipment used, the anesthetic and non-anesthetic drugs used, the clinical and paraclinical neurological and cardio-respiratory parameters and the nature of the complications following anaesthetic induction will be collected up to the 10th post-induction minute.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years' old
* Procedure requiring general anesthesia with oro or nasotracheal intubation
* Anesthetic management with indication of rapid sequence induction
* No objection after oral and written information to the patient

Exclusion Criteria:

* Age < 18 years' old
* Impossible intubation planned
* Preoperative respiratory distress (SpO2 < 90% in ambient air)
* Preoperative shock (MBP≤ 65 mmHg or vasopressive amines)
* Preoperative coma defined by a Glasgow score ≤ 12/15
* Patient in cardiopulmonary arrest
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients for whom rapid sequence anesthetic induction has been retained in the operating room and for whom no opposition has been obtained during the anesthesia consultation will be included consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a major haemodynamic disorder | Within the first 10 minutes after induction of anesthesia
  MBP ≤ 50 mmHg (or ≤ 40% of the reference value) and/or ≥ 110 mmHg and/or occurrence of a sustained arrhythmia (> 1 min) not present at induction and/or cardiac arrest

SECONDARY OUTCOMES:
Clinical pre-anesthesic assessment of the risk of a full stomach | From 6 hours before induction of anesthesia until the beginning of the preoxygenation for the rapid sequence induction procedure
  - percentage of clinical and/or imaging endpoints in favor of a full stomach
Pre-anesthetic assessment of the risk of a full stomach | From 6 hours before induction of anesthesia until the beginning of the preoxygenation for the rapid sequence induction procedure
  - percentage of gastric ultrasound use
Assessment of the risk of a full stomach | From 6 hours before induction of anesthesia until the beginning of the preoxygenation for the rapid sequence induction procedure
  - percentage of presence and use of the Nasogastric Tube
Team involved in the rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - average number of individuals in the room participating in the performance of SRI
Preparation for rapide sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - Percentage of patients in supine position
Use of morphine for rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - percentage of use of morphine derivative prior to airway securisation
Induction therapeutics for rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - percentage of use of each of the following hypnotics: propofol, ketamine, thiopental, etomidate, midazolam, sevoflurane
Use of curare for rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - percentage of use of a curare
Use of vasopressive amine for rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - percentage and median dosage of vasopressive amine use for the prevention of low blood pressure
Use of filling solution for rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - percentage and median volume of use of a preventive vascular filling solution
Airway management for rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - type of preoxygenation
Operator qualification for rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - percentages of first operator with a medical degree, of trained nurses, and of medical resident performing the rapid sequence induction technique
Laryngoscopy for rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - percentage of use of a video laryngoscope as a 1st intention
Medical device used for rapid sequence induction technique | Within the first 10 minutes after induction of anesthesia
  - percentage of mandrel use at the first laryngoscopy
MBP complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - percentage of episode of MBP ≤ at 50 mmHg (or ≤ 40% of the baseline)
Tension complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - percentage of episode of MBP ≥ 110 mmHg
Rythmal complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - sustained arrhythmia (> 1 minute) not present at induction
Cardiac complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - cardiac arrest
Intubation complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - percentage of intubations that required more than one laryngoscopy
Low tension-related complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - percentage and median dosage of use of a vasopressive amine required for the treatment of low blood pressure (defined as a SBP < 80 mmHg)
High tension-related complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - percentage of use of an antihypertensive drug or sedation-analgesia bolus for the treatment of high blood pressure (defined as SBP > 160 mmHg)
Respiratory complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - percentage of respiratory complication defined by Spo2 < 90% or the need for manual reventilation
Anaphylactic complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - percentage of Grade I, II, III or IV anaphylactic reaction
Inhalation complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - percentage of gastric fluid inhalation defined by the presence of non-salivary fluid or supraglottic solids during laryngoscopy
Immediate complications of ISR (< 10 minutes) | Within the first 10 minutes after induction of anesthesia
  - percentage of intraoperative deaths

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Grillot, MD, Study Director — Nantes University Hospital
Locations (42):
- France (42):
  - Clinique Victor Pauchet, Amiens
  - Hospital, Arcachon
  - Hospital, Armentières
  - Hôpital Privé Arras les Bonnettes, Arras
  - University Hospital, Brest
  - University Hospital, Caen
  - Centre Hospitalier Intercommunal, Castres
  - University Hospital, Clermont-Ferrand
  - CHD Vendée, La Roche-sur-Yon
  - University Hospital, Lille
  - Hospital, Lorient
  - Centre Léon Bérard, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Saint Joseph Saint Luc Hospital, Lyon
  - University Hopital - Edouard Herriot, Lyon
  - University Hospital - Sud, Lyon
  - Hospital, Mont-de-Marsan
  - Hospital, Montargis
  - University Hospital, Nantes
  - University Hospital - Pasteur, Nice
  - Bichat Hospital - APHP, Paris
  - Hopital Lariboisiere - APHP, Paris
  - Hopital Pitié Salpetriere - APHP, Paris
  - Hopital Saint Louis, Lariboisiere, Fernand Widal - APHP, Paris
  - Hôpital Tenon - APHP, Paris
  - University Hospital, Poitiers
  - Clinique de la Sagesse, Rennes
  - Hospital, Rodez
  - Yves Le Foll Hospital, Saint-Brieuc
  - University Hospital La Réunion - Site Nord, Saint-Denis
  - University Hospital La Réunion - site Ouest, Saint-Paul
  - Groupe Hospitalier Seclin Carvin, Seclin
  - Centre Clinical - Angoulême, Soyaux
  - Hospital, St-Malo
  - Clinique Rhéna, Strasbourg
  - University Hospital - Hautepierre, Strasbourg
  - Hôpitaux du Leman, Thonon-les-Bains
  - Centre hospitalier intercommunal, Toulon
  - University Hospital - Rangueil, Toulouse
  - Hospital, Valenciennes
  - Institut Gustave Roussy, Villejuif
  - Clinique de Villeneuve Saint Georges, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: Undecided